CLINICAL TRIAL: NCT03789019
Title: Estimation of the Optimal Treatment Duration and Cumulative Dose of BP-C1 in Breast Cancer Patients With Distant Metastases: a Dose-response Study (IC)
Brief Title: BP-C1 Monotherapy in Patients With Metastatic Breast Cancer Cancer: Estimation of Optimal Duration of Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meabco A/S (Industry)
Collaborators: Meddoc (Other); Norwegian University of Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMC2011-02
Record Dates: First submitted 2018-12-23; First posted 2018-12-28 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Metastatic Breast Cancer; Stage IV Breast Cancer
Keywords: BP-C1; Cis-coordinated complexes of platinum(II) with polymer of benzene polycarboxylic acids derived from lignin; Benzene polycarboxylic acids complex with cis-diammineplatinum( II); Metastatic Breast Cancer; Platinum analogue; Metronomic chemotherapy; Breast cancer; Cisplatin; cis-diammineplatinum(II) complexed with a polymer containing benzene polycarboxylic acids derived from lignin
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BP-C1 (Experimental): Dose-response part: patients who have completed the first 32-day treatment period with BP-C1 under Protocol BMC2011-1/Protocol MBC-BPC1/IIB or Protocol BMC2012-4, and having a maximum of "moderate" toxicity at the end of treatment are offered to continue in the second 32-day treatment period with BP-C1 under the protocol BMC2011-02. Patients completing 64-day treatment period with BP-C1 will be followed up for 28 days.
  Follow-up study: the patients will be given BP-C1 as long as they obtain benefit from the treatment (i.e. until disease progression or increase in toxicity not above "moderate" grade).
  Interventions: Drug: BP-C1

INTERVENTIONS:
Drug: BP-C1 — BP-C1, 0.05% solution for injection; doses: 0.035 mg/kg body weight (0.07 mL/kg) intramuscularly once daily for 32 consecutive days
  Other Names: Cis-coordinated complexes of platinum(II) with polymer of benzene polycarboxylic acids derived from lignin; Cis-diammineplatinum(II) complexed with a polymer containing benzene polycarboxylic acids derived from lignin

SUMMARY:
The purpose of this study is to establish an optimal treatment duration and tolerable cumulative dose for BP-C1 in the treatment of metastatic breast cancer patients who had previously undergone at least three lines of chemotherapy.

DETAILED DESCRIPTION:
BP-C1, solution for injection 0.05%, is currently being developed for treatment of patients with metastatic breast cancer with palliative intent. Active substance of the product, which is a novel platinum-containing anticancer agent developed for intramuscular administration, is cis-diammineplatinum(II) complexed with a polymer containing benzene polycarboxylic acids derived from lignin. The amphiphilic characteristics of the polymer have resulted in a product with clear and significantly altered and improved properties compared to other platinum analogues, e.g. cisplatin, carboplatin and oxaliplatin.

BP-C1 preserves antitumour activity of its predecessors (e.g. cisplatin and carboplatin), additionally offering the following advantages that ensure favourable outcome of treatment of metastatic breast cancer patients:

* injectable solution (intramuscular) does not cause injection site reactions;
* can be administered at home by a nurse or a patient;
* has an improved pharmacokinetic profile;
* demonstrates efficacy comparable to cisplatin and much higher than carboplatin (in-vitro; in-vivo data);
* exerts an additional immunomodulatory activity.

This study is an open-label, non-randomised, single-group, multi-centre study with a sequential safety design. The study consists of two parts: dose-response part and follow-up study.

Dose-response part: Patients who have completed the first 32-day treatment period with BP-C1 from Day 1 to Day 32 under Protocol BMC2011-1/Protocol MBC-BPC1/IIB or Protocol BMC2012-4, and having a maximum of "moderate" toxicity at the end of treatment are offered to continue in the second 32-day treatment period with BP-C1 from Day 33 to Day 64 under protocol BMC2011-02. Patients completing 64-day treatment period with BP-C1 will be followed up for 28 days.

Follow-up study: After 28-day follow-up period the patients without disease progression and without an increase in toxicity are offered to participate in the follow-up study. During the follow-up study the patients will be given BP-C1 as long as they obtain benefit from the treatment (i.e. until disease progression or increase in toxicity not above "moderate" grade).

ELIGIBILITY:
Inclusion Criteria:

Female patients who have completed 32-day treatment with BP-C1 (under protocols BMC2011-1, MBC-BPC1/IIA, BMC2012-4), having increase in toxicity not above moderate level, and having no progression of the disease. In accordance with inclusion criteria checked in the studies BMC2011-1, MBC-BPC1/IIA, or BMC2012-4, the patients are between 18 and 80 years with metastatic breast cancer (stage IV), had previously underwent at least third line chemotherapy, and have an expected survival time of at least 3 months.

Exclusion Criteria:

* Severe or life-threatening increase in toxicity after preceding 32-day treatment with BP-C1.
* Abnormal liver function classified as total bilirubin >34 μmol/L or ALAT > 3 times of the upper limit of normal (ULN). In case of metastases in the liver, the ALAT limit for exclusion is set to 5хULN.
* Abnormal kidney function defined by serum creatinine >120 μmol/L.
* Abnormal coagulation capacity defined by the relative arbitrary concentration of coagulation factors 2,7,10 <0.70 or international normalised ratio (INR) >1.5.
* Verified metastases to the brain.
* Synchronous cancer except for non-melanoma skin cancer and early stage of cervical cancer.
* Abnormal hematology status defined by hemoglobin < 9.0 g/dL, platelet count <100,000/mm^3 or leucocytes < 3 x 10^9/L.
* Clinically significant abnormal ECG.
* Karnofsky performance status score <60%.
* Pregnant or breast-feeding women.
* Women of fertile age who do not want to be tested for possible pregnancy.
* Fertile female who do not want to use safe protection against pregnancy, starting one month before the start of the study treatment and lasting at least six weeks after.
* Uncontrolled bacterial, viral, fungal or parasite infection.
* Under systemic treatment with corticosteroids or other immunosuppressive drugs in the last 3 weeks before start of the trial treatment.
* Participating in another clinical trial with pharmaceuticals in the last six weeks before start of this trial treatment.
* Not able to understand information.
* Not willing or not able to give written consent to participate in the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-02-22 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2016-07-29 (Actual)

PRIMARY OUTCOMES:
Sum Common Toxicity Criteria score (Sum CTC score) | baseline to Day 64 of treatment period
  Toxicity will be assessed according to National Cancer Institute Common Toxicity Criteria version 2.0 (CTC v2.0). The CTC v2.0 is divided in 15 toxicity categories (variables); each category is divided by corresponding sub-variables. Each sub-variable is measured on five-point fixed scale from 0 to 4: 0-none, 1-mild, 2-moderate, 3-severe, 4-life-threatening. However, in this trial each sub-variable will be measured on modified fixed scale from 1 to 4: 1-none or mild, 2-moderate, 3-severe, 4-life-threatening. The classification of each toxicity variable will be judged based on the largest observed value for its sub-variables. The Sum CTC score will be calculated by taking the sum of each variable across all categories.
Maximum Common Toxicity Criteria score (Maximum CTC score) | baseline to Day 64 of treatment period
  Toxicity will be assessed according to National Cancer Institute Common Toxicity Criteria version 2.0 (CTC v2.0). The CTC v2.0 is divided in 15 toxicity categories (variables); each category is divided by corresponding sub-variables. Each sub-variable is measured on five-point fixed scale from 0 to 4: 0-none, 1-mild, 2-moderate, 3-severe, 4-life-threatening. However, in this trial each sub-variable will be measured on modified fixed scale from 1 to 4: 1-none or mild, 2-moderate, 3-severe, 4-life-threatening. The classification of each toxicity variable will be judged based on the largest observed value for its sub-variables. The Maximum CTC score will be calculated by taking the maximum value among all variables across all categories.

SECONDARY OUTCOMES:
Change (%) in the sum of diameters of target lesions | baseline to Day 64 of treatment period
  Diameter of target lesions will be measured by computer tomography (CT) with contrasting using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Treatment response | baseline to Day 64 of treatment period
  In accordance with RECIST v1.1 the treatment response will be classified as 'complete response', 'partial response', 'stable disease' or 'progressive disease': Complete response (CR): disappearance of all target lesions. Partial response (PR): at least 30% decrease in the sum of longest diameters of target lesions, taking as reference the baseline sum of diameters. Progressive disease (PD): at least 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum might also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions will also be considered progression. Stable disease (SD): neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Karnofsky Performance Status score (KPS score) | baseline to Day 64 of treatment period
  KPS score will give an outcome with 11 grades, starting as normal status without complaints and evidence of disease as the best (KPS score = 100) and the dead status as the lowest (KPS score = 0)
Changes in sub-scores of the three major scales of general quality of life questionnaire (EORTC QLQ-C30) | baseline to Day 64 of treatment period
  Quality of life sub-scores will be obtained by general cancer questionnaire EORTC QLQ-C30. EORTC QLQ-C30 consists of 30 questions generally related to cancer. The questionnaire will be self-administered and will be given in patient's mother tongue. EORTC QLQ-C30 (version 3) is divided in the 3 major scales that will be presented as 15 sub-scores: i) global health status; ii) functional scale (physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning); iii) symptom scale/item(fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea, financial difficulties). Range of functional scale is 0-100 (high values are "better"). Range of symptom scale is 0-100 (low values are "better").
Changes in sub-scores of the specific quality of life questionnaire (EORTC QLQ-BR23) | baseline to Day 64 of treatment period
  Quality of life sub-scores will be obtained by specific breast cancer questionnaire EORTC QLQ-BR23. EORTC QLQ-BR-23 consists of 23 questions related to breast cancer. The questionnaire will be self-administered and will be given in patient's mother tongue. EORTC QLQ-BR23 is divided in 2 scales that will be presented as 8 sub-scores: i) functional scale (body image, sexual functioning, sexual enjoyment, future perspective); ii) symptom scale/item (systemic therapy side effect, breast symptom, arm symptom, upset by hair loss). Range of functional scale is 0-100 (high values are "better"). Range of symptom scale is 0-100 (low values are "better").
Number of registered adverse events | baseline to Day 28 of follow-up period
  Adverse events (AEs) will be coded according to the MedDRA (version 16.1E). AEs will be systemized by system organ class and by preferred term. AEs will be analyzed by severity, seriousness and relatedness to the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Henning Arboe, Study Chair — Meabco A/S
Locations (7):
- Russia (3):
  - Russian Oncological Research Centre n.a. N.N. Blokhin, Russian Academy of Medical Science (RAMS), Moscow
  - Leningrad Regional Oncological Centre, Saint Petersburg
  - St. Petersburg State Budgetary Health Organization, City Clinical Oncology Dispensary, Saint Petersburg
- Thailand (4):
  - Siriraj Hospital, Mahidol University, Bangkok
  - Lampang Cancer Hospital, Lampang
  - Ubon Ratchanthani Cancer Hospital, Ubon Ratchathani
  - Udon Thani Cancer Hospital, Udon Thani

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Larsen S, Butthongkomvong K, Manikhas A, Trishkina E, Poddubuskaya E, Matrosova M, Srimuninnimit V, Lindkaer-Jensen S. BP-C1 in the treatment of patients with stage IV breast cancer: a randomized, double-blind, placebo-controlled multicenter study and an additional open-label treatment phase. Breast Cancer (Dove Med Press). 2014 Nov 27;6:179-89. doi: 10.2147/BCTT.S71781. eCollection 2014. PMID 25473312
- [Result] Lindkaer-Jensen S, Larsen S, Habib-Lindkaer-Jensen N, Fagertun HE. Positive effects on hematological and biochemical imbalances in patients with metastatic breast cancer stage IV, of BP-C1, a new anticancer substance. Drug Des Devel Ther. 2015 Mar 13;9:1481-90. doi: 10.2147/DDDT.S80451. eCollection 2015. PMID 25792808